CLINICAL TRIAL: NCT05654415
Title: Efficacy of Melatony Versus Sleep Deprivation for EEG Recordings in Sleep: a Randomized Crossed-over Study in Pediatric Patients With Epilepsy
Brief Title: Melatonin vs Sleep Deprivation for Nap EEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MLT2022
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Epilepsy
Keywords: Oral melatonin; Sleep deprivation; Nap EEG recordings; Time to fall asleep
MeSH Terms: conditions — Epilepsy; Sleep Deprivation | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The patients will be subjected to two EEG recordings: in one they will receive the melatonin solution (5 mg), in the 'other they will undergo only partial sleep deprivation (about 50% of physiological sleep).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deprivation group (Experimental): Sleep deprivation of 50% of physiological sleep
  Interventions: Other: Deprivation
- Melatonin group (Experimental): Melatonin oral solution 5 mg 30 minutes before EEG performing
  Interventions: Other: Melatonin

INTERVENTIONS:
Other: Melatonin — Each enrolled patient will be subjected to two nap EEG recordings receiving in one occasion the melatonin-based solution under study at a dosage of 5 mg
  Arms: Melatonin group
Other: Deprivation — Each enrolled patient will be subjected to two nap EEG recordings,in one they will be subjected to sleep deprivation
  Arms: Deprivation group

SUMMARY:
In the pediatric population, electroencephalographic (EEG) recordings are frequently performed in sleep, as it reduces the amount of artifacts and might activate epileptiform discharges. To date, no agreed-upon guidelines are available for hypno-induction for EEG recordings . Among the strategies used, the most commonly used are sleep deprivation, either total or partial, and the use of melatonin, alone or in combination. The investigators proposed a study aiming at evaluating the efficacy of a melatonin-based solution for sleep induction during EEG video recording VS sleep deprivation.

In a randomized, crossover study, 30 pediatric patients (aged 4-10 years) will be subjected to two EEG recordings: in one they will receive the melatonin solution (5 mg), in the other they undergo only partial sleep deprivation (about 50% of physiological sleep). The primary endpoint of the study is represented by the time to fall asleep, secondary objectives are represented by frequency of epileptiform discharges, presence/absence of epileptic seizures, In addition, the levels of 6-sulfatoxymelatonina, the primary metabolite of melatonin in saliva and urine, will be determined with a validated LC-MS method.

DETAILED DESCRIPTION:
Background: Electroencephalographic recording is essential in children with suspected or diagnosed epilepsy. Due to difficulties in obtaining a reliable EEG, in pediatric patients electroencephalographic recordings are often performed during sleep in order to reduce the number of artefacts connected to movements and to activate epileptic discharges. To date, there are no shared guidelines about hypno-induction. Most of hypnotic drugs such as benzodiazepines and barbiturates are known to alter EEG registration, by changing background activity or epileptiform activities. Clinicians often aim to induce sleep by total or partial sleep deprivation. A recent survey assessing strategies used by various centers in Italy highlights that there is a great heterogeneous approach to obtain hypno-induction. Among sleep-inductive interventions, the use of melatonin is the most common alone or in combination with sleep-deprivation. Melatonin is a hormone (N-acetylmethoxytryptamine), produced by the pineal gland, whose secretion is regulated by the suprachiasmatic nucleus of the hypothalamus and which is able to regulate circadian rhythms. An open-lable study evaluated the role of melatonin on the EEG recordings (artefacts, anomalies) and its efficacy in inducing sleep in 50 children with epilepsy or with neurodevelopmental disorders. This study demonstrates that melatonin is not more effective than sleep deprivation in hypno-induction, without modifying the EEG pattern. Furthermore, melatonin is equally efficient as partial sleep deprivation in inducing sleep and does not affect the occurrence of epileptic discharges in the EEG recording. Another recent study combined sleep deprivation and melatonin revealing the greater effectiveness of the combination of the two methods against the use of them individually. However, this study was not randomized. Moreover, there is no clear consensus about when and in which doses melatonin should be administrated in children: doses vary between different studies ranging from 2 to 20 mg.

From these observations it is clear, therefore, that the role of melatonin is strategic in hypno-induction and no cases of toxicity or adverse effects in the short and long term deriving from the use of melatonin are known in the literature. The aim of this randomized study is to determine non-inferiority of melatonin 5 mg against sleep deprivation in inducing sleep in a cohort of children and adolescents with epilepsy and to determine if melatonin could affect the frequency of epileptic discharges or clinically detectable epileptic seizures during nap EEG recordings. Furthermore, the investigators try to indicate an adequate dose for melatonin for hypno-induction. Moreover, the levels of 6-sulfatoxymelatonina, the primary metabolite of melatonin in saliva and urine, will be determined with a validated LC-MS method to detect a possible correlation between sleep induction and melatonin metabolism.

Each enrolled patient will be subjected to two nap EEG recordings receiving in one the melatonin-based solution under study at a dosage of 5 mg, in the other they will be subjected to sleep deprivation (defined as 50% of physiological sleep). The electroencephalographic recordings with video and polygraphy in siesta at the same time, will be performed at a time distance of 1-3 months.

The study is open label and therefore no masking method is used. In order to minimize the bias deriving from the open label situation, the calculation of the time to fall asleep is based on objective EEG parameters (disappearance of the background rhythm of the alpha band on the posterior regions and appearance of the physiological hypnic figures, characteristics of the N1 phase of non-REM sleep), as well as the calculation of the frequency of epileptic anomalies which occurs through the use of special instrumentation (so-called "tip counter tool", an automatic tool for detecting epileptiform anomalies on the electroencephalographic trace ).

In addition, the levels of 6-sulfatoxymelatonina, the primary metabolite of melatonin in saliva and urine, will be determined with a validated LC-MS method.

Duration of the study: 52 weeks Duration of enrollment: 36 weeks

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with epilepsy aged between 4 and 10 years with normal psychomotor development and IQ> 70;
* stable seizure frequency in the 3 months preceding the enrollment ;
* stable anti-seizure medications in the 3 months preceding the enrollment;
* written informed consent from the legal representative.

Exclusion Criteria:

* subjects diagnosed with obstructive sleep apnea or other sleep disorders;
* history of neurodevelopmental disorders;
* concomitant use of hypnotics, stimulants, systemic corticosteroids or other immunosuppressants;
* concomitant daily use of melatonin;
* any conditions which, in the investigator's judgment, would compromise the achievement of the study objectives;
* refusal to sign the informed consent from the legal representative.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time elapsed (in seconds) from the starting of the EEG and beginning of sleep stages at EEG recording with melatonin | From 0 seconds to 1.5 hours
  Disappearance of the background rhythm of the alpha band on the posterior regions and appearance of the physiological hypnic figures, characteristics of the N1 phase of non-REM sleep
Time elapsed (in seconds) from the starting of the EEG and beginning of sleep stages at EEG recording with deprivation | From 0 seconds to 1.5 hours
  Disappearance of the background rhythm of the alpha band on the posterior regions and appearance of the physiological hypnic figures, characteristics of the N1 phase of non-REM sleep

SECONDARY OUTCOMES:
Frequency of epileptic anomalies | From 0 seconds to 1.5 hours
  Anomalies which occurs through the use of special instrumentation (so-called "tip counter tool", an automatic tool for detecting epileptiform anomalies on the electroencephalographic trace
Clinically detectable seizures | From 0 seconds to 1.5 hours
  Presence/absence ofseizures
Levels of 6-sulfatoxymelatonina | 120 minutes after oral melatonin solution
  Determination of the levels of the primary metabolite of melatonin in saliva and urine, with a validated LC-MS method

CONTACTS AND LOCATIONS:
Overall Officials: Valentina De Giorgis, MD, Principal Investigator — Child and Adolescent Epileptology Center
Locations (1):
- Child and Adolescent Epileptology Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alix JJP, Kandler RH, Pang C, Stavroulakis T, Catania S. Sleep deprivation and melatonin for inducing sleep in paediatric electroencephalography: a prospective multicentre service evaluation. Dev Med Child Neurol. 2019 Feb;61(2):181-185. doi: 10.1111/dmcn.13973. Epub 2018 Jul 20. PMID 30028504
- [Background] Eisermann M, Kaminska A, Berdougo B, Brunet ML. Melatonin: experience in its use for recording sleep EEG in children and review of the literature. Neuropediatrics. 2010 Aug;41(4):163-6. doi: 10.1055/s-0030-1267920. Epub 2010 Nov 17. PMID 21086220
- [Background] Gasparini S, Sueri C, Ascoli M, Cianci V, Cavalli SM, Ferrigno G, Belcastro V, Aguglia U, Ferlazzo E; Epilepsy Study Group of the Italian Neurological Society. Need for a standardized technique of nap EEG recordings: results of a national online survey in Italy. Neurol Sci. 2018 Nov;39(11):1911-1915. doi: 10.1007/s10072-018-3525-9. Epub 2018 Aug 23. PMID 30140986
- [Background] Gustafsson G, Brostrom A, Ulander M, Vrethem M, Svanborg E. Occurrence of epileptiform discharges and sleep during EEG recordings in children after melatonin intake versus sleep-deprivation. Clin Neurophysiol. 2015 Aug;126(8):1493-7. doi: 10.1016/j.clinph.2014.10.015. Epub 2014 Oct 18. PMID 25453612
- [Background] Jain SV, Horn PS, Simakajornboon N, Beebe DW, Holland K, Byars AW, Glauser TA. Melatonin improves sleep in children with epilepsy: a randomized, double-blind, crossover study. Sleep Med. 2015 May;16(5):637-44. doi: 10.1016/j.sleep.2015.01.005. Epub 2015 Jan 21. PMID 25862116
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Liamsuwan S, Grattan-Smith P, Fagan E, Bleasel A, Antony J. The value of partial sleep deprivation as a routine measure in pediatric electroencephalography. J Child Neurol. 2000 Jan;15(1):26-9. doi: 10.1177/088307380001500106. PMID 10641606
- [Background] Sander J, Shamdeen MG, Gottschling S, Gortner L, Graber S, Meyer S. Melatonin does not influence sleep deprivation electroencephalogram recordings in children. Eur J Pediatr. 2012 Apr;171(4):675-9. doi: 10.1007/s00431-011-1640-1. Epub 2011 Nov 29. PMID 22124712
- [Background] Smith SJ. EEG in the diagnosis, classification, and management of patients with epilepsy. J Neurol Neurosurg Psychiatry. 2005 Jun;76 Suppl 2(Suppl 2):ii2-7. doi: 10.1136/jnnp.2005.069245. No abstract available. PMID 15961864
- [Background] Wassmer E, Quinn E, Whitehouse W, Seri S. Melatonin as a sleep inductor for electroencephalogram recordings in children. Clin Neurophysiol. 2001 Apr;112(4):683-5. doi: 10.1016/s1388-2457(00)00554-x. PMID 11275541
- [Background] Wassmer E, Carter PF, Quinn E, McLean N, Welsh G, Seri S, Whitehouse WP. Melatonin is useful for recording sleep EEGs: a prospective audit of outcome. Dev Med Child Neurol. 2001 Nov;43(11):735-8. doi: 10.1017/s0012162201001347. PMID 11730146